CLINICAL TRIAL: NCT05502718
Title: Evaluation of the Effect of Personalized Exercise Program on Clinical Findings and Quality of Life of Patients With Cervical Dystonia Who Received Botulinum Toxin Type A Injection
Brief Title: Exercise Program for Patients With Cervical Dystonia Who Are Treated With Botulinum Toxin Type A
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Şehim Kutlay (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Şehim Kutlay, Prof.Dr., Ankara University
Organization: Ankara University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I05-279-22
Record Dates: First submitted 2022-07-28; First posted 2022-08-16 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Dystonia, Cervical
Keywords: Botulinum Toxin Type A; Exercise; Quality of Life
MeSH Terms: conditions — Torticollis; Motor Activity | interventions — Respiration

STUDY DESIGN:
Intervention Model Description: Patients with cervical dystonia who received botulinum toxin type A injection will be divided into study group and control group.The patients in the study group will be given stretching, strengthening, breathing and rhythmic coordination exercises for the muscles involved. (Personalized exercise program) In the control group, only breathing and rhythmic coordination exercises will be given and the two groups will be compared.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group (Active Comparator): The patients in the study group will be given stretching, strengthening, breathing and rhythmic coordination exercises for the muscles involved. (Personalized exercise program)
  Interventions: Other: Stretching and Strengthening Exercises; Other: Breathing and Rhythmic Coordination Exercises
- Control Group (Placebo Comparator): The patients in the control group will be given only breathing and rhythmic coordination exercises.
  Interventions: Other: Breathing and Rhythmic Coordination Exercises

INTERVENTIONS:
Other: Stretching and Strengthening Exercises — The patients in the study group will be given exercise videos. These exercise videos will be selected in accordance with the patient's cervical dystonia type (Torticollis, laterocollis, retrocollis, anterocollis). During the exercises, stretching exercises will be applied to the muscle groups that cause dystonia, and isometric strengthening exercises will be applied to the contralateral muscle groups. Videos including breathing exercises and rhythmic coordination exercises will also be given to all patients in the study and control groups. Patients will be asked to do these exercises for 10 repetitions, three times a day, five days a week. Patients will be asked to mark after each exercise on the exercise chart prepared to determine continuity and compliance with exercise. Patients will be called and followed up on a weekly basis with the exercise chart given to the patients and by telephone.
  Arms: Study Group
Other: Breathing and Rhythmic Coordination Exercises — The patients in the study group will be given exercise videos prepared in the Department of Physical Medicine and Rehabilitation of Ankara University Faculty of Medicine. . Videos including breathing exercises and rhythmic coordination exercises will also be given to all patients in the study and control groups. Patients will be asked to do these exercises for 10 repetitions, three times a day, five days a week.

SUMMARY:
Dystonia is involuntary movements characterized by posture abnormalities or repetitive movements as a result of continuous or intermittent simultaneous contraction of opposing muscle groups. Dystonic movements are twisted and twisted in a certain pattern. Dystonia is named in different ways according to its distribution in the body. Cervical dystonia is the most common form of regional dystonia and can be defined as involuntary movements of the head in normal upright posture.Cervical dystonia has different names according to the posture of the neck (torticollis, laterocollis, anterocollis and retrocollis). These different postures can be seen individually as well as together.Pain in cervical dystonia is seen in approximately 70% of patients, and this condition is closely related to involuntary contractions of neck muscles and neck posture disorder. Fatigue, anxiety, unhappiness, decreased self-efficacy and limitation in daily living activities due to decreased neck movements are the main causes of disability in patients with cervical dystonia. The first-line treatment of cervical dystonia consists of injecting botulinum toxin type A into the relevant muscles to alleviate these complaints.There is increasing evidence that range of motion, stretching, and relaxation exercises, in addition to botulinum toxin therapy, have beneficial effects on pain and disability in patients with cervical dystonia.In this study, patients with cervical dystonia who received botulinum toxin type A injection will be divided into study group and control group.The patients in the study group will be given stretching, strengthening, breathing and rhythmic coordination exercises for the muscles involved. (Personalized exercise program) In the control group, only breathing and rhythmic coordination exercises will be given and the two groups will be compared.Thus, it is aimed to investigate the effect of a personalized exercise program on clinical findings and the patient's quality of life.

DETAILED DESCRIPTION:
Restriction of neck movements, pain, decrease in participation in activities of daily living and decrease in quality of life are common complaints in patients with cervical dystonia.Botulinum toxin injections are indisputably one of the most preferred methods in the treatment.There are debates about the contribution of exercise to treatment in these patients with functional limitation and pain.It is thought that the exercise program after botulinum toxin injection may be effective in reducing the patient's complaints and increasing the quality of life. Exercise programs can be planned as supervised or self-executed. However, although the effectiveness of supervised exercises is higher due to better patient compliance, it also brings a burden to both patients and the health system as it requires the patient to come to a center.

In this study, patients with cervical dystonia who received botulinum toxin type A injection will be divided into study group and control group.The patients in the study group will be given stretching, strengthening, breathing and rhythmic coordination exercises for the muscles involved. (Personalized exercise program) In the control group, only breathing and rhythmic coordination exercises will be given and the two groups will be compared.Thus, it is aimed to investigate the effect of a personalized exercise program on clinical findings and the patient's quality of life.

Dystonia is involuntary movements characterized by postural abnormalities or repetitive movements as a result of continuous or intermittent simultaneous contractions of opposing muscle groups.Dystonic movements are twisted and twisted in a certain pattern. Dystonia can be focal, segmental, multifocal, generalized or hemidystonia according to its distribution in the body.It is classified as primary (idiopathic) and secondary according to the etiology. Cervical dystonia is the most common form of focal dystonia and can be defined as involuntary postural movements of the head in normal upright posture.There are different types of cervical dystonia such as torticollis, laterocollis, anterocollis and retrocollis. These forms can be seen individually as well as in combination. The dystonic position can be intermittent or continuous. It may also be accompanied by tremor.Idiopathic cervical dystonia has a prevalence of 5-9 per 100,000. The mean age of onset is 42 years, and it is seen in relatively young individuals. It is seen 1.5-1.9 times more in women than in men. Pain is seen in approximately 70% of patients and is closely related to involuntary contractions of neck muscles and impaired neck posture. Fatigue, anxiety, depression, decreased self-efficacy and limitation in daily living activities due to limitation in neck movements are the main causes of disability in patients with cervical dystonia. Before starting treatment in patients followed up with a diagnosis of dystonia, it is necessary to make sure that the distinction between primary and secondary dystonia is made correctly. Because secondary dystonias can occur due to many reasons and elimination of the cause constitutes the first step of treatment.Discontinuation of treatment in drug-induced dystonias, and treatment of the disease primarily in metabolic diseases can be given as examples. With symptomatic treatment in cervical dystonia, it is aimed to improve the quality of life by reducing symptoms such as muscle contractions, abnormal head and neck posture, pain and tremor, and to prevent secondary complications such as myelopathy, radiculopathy and dysphagia. Treatment options in cervical dystonia can be examined under three headings. These are pharmacological treatments, surgical treatments and chemodenervation (botulinum toxin injection application) options. In some cases, it may be necessary to combine these options.

Patients who meet the inclusion criteria after botulinum toxin injection application due to cervical dystonia in the Department of Neurology, Department of Neurology, Ankara University will be invited to the study. Before the study, patients will be asked to review the informed consent form and give their consent to the study. Socio-demographic information (name-surname, gender, age, education level, marital status, occupation, contact information, file numbers) of all patients who accepted to participate in the study will be recorded. Additional diseases, medications used, total number of botulinum toxin administered for cervical dystonia, date of diagnosis and symptoms of cervical dystonia will be questioned in the history of the patients. After this stage, patients will be randomized into two groups as study and control groups. Patients in both the study and control groups will consist of patients with a diagnosis of cervical dystonia and botulinum toxin injections. The patients in the study group will be given exercise videos prepared in the Department of Physical Medicine and Rehabilitation of Ankara University Faculty of Medicine. These exercise videos will be selected in accordance with the patient's cervical dystonia type (Torticollis, laterocollis, retrocollis, anterocollis). During the exercises, stretching exercises will be applied to the muscle groups that cause dystonia, and isometric strengthening exercises will be applied to the contralateral muscle groups. Videos including breathing exercises and rhythmic coordination exercises will also be given to all patients in the study and control groups. Patients will be asked to do these exercises for 10 repetitions, three times a day, five days a week. Patients will be asked to mark after each exercise on the exercise chart prepared to determine continuity and compliance with exercise. Patients will be called and followed up on a weekly basis with the exercise chart given to the patients and by telephone.

The primary outcome measure will be a change from baseline of at least 5 units in the torticollis pain scale, a subscale of the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS), with 12 weeks of exercise.

The calculation of the sample size will be based on the primary dependent variable.

Using the G-Power program version 3.1.9.2, an alpha error of 5%, a ß error of 20%, and a patient loss rate of 20% were determined, and 17 volunteers were recruited to the study group and control group at 80% power.

Statistical Package for the Social Sciences(SPSS) 11.5 package program will be used in the evaluation of the data.

Frequency (percentage) for the variables obtained by counting, mean (standard deviation) for the variables obtained by measurement will be given as descriptive statistics.

In intergroup comparisons, t-test will be used in independent groups for variables obtained by measurement, and chi-square test will be used for variables obtained by counting.

Analysis of variance will be used in repeated measurements to examine the trend of time-dependent change in groups.

p<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years old
* Completion of Informed Signed Consent Form
* Diagnosis of cervical dystonia by neurology
* Botulinum toxin injection for cervical dystonia in Ankara University Faculty of Medicine Neurology Department Movement Disorders Outpatient Clinic
* To have the necessary infrastructure to watch the prepared exercise videos on computers, phones, tablets.

Exclusion Criteria:

* Cardiovascular, systemic or musculoskeletal problems that prevent participation in the exercise program
* Presence of dementia/cognitive disorder or symptomatic psychiatric disease, which was previously diagnosed or detected during the anamnesis process, preventing participation in the program
* Failure to approve the Informed Signed Consent Form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-09-17 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Toronto Western Spasmodic Torticollis Rating Scale Subscale Torticollis Pain Scale (0-20) | 0-6-12. Week
  A change of at least 5 units from baseline in the torticollis pain scale (0-20), which is a subscale of the Toronto Western Spasmodic Torticollis Rating Scale, after 12 weeks of exercise application. (Higher scores mean a worse outcome.)

SECONDARY OUTCOMES:
Toronto Western Spasmodic Torticollis Rating Scale Subscale Disability Scale(0-30) | 0-6-12. Week
  Detection of improvement from baseline in the disability subscale(0-30) of the Toronto Western Spasmodic Torticollis Scale (Higher scores mean a worse outcome.)
Toronto Western Spasmodic Torticollis Rating Scale Subscale Severity Scale (0-35) | 0-6-12. Week
  Detection of improvement from baseline in the severity subscale(0-35) of the Toronto Western Spasmodic Torticollis Scale (Higher scores mean a worse outcome.)
Craniocervical dystonia questionnaire (0-100) | 0-6-12. Week
  Improvement in quality of life as assessed by the Craniocervical dystonia questionnaire (0-100) (Higher scores mean a worse outcome.)

CONTACTS AND LOCATIONS:
Overall Officials: Sehim Sehim, Study Director — sehim.kutlay@gmail.com
Locations (1):
- Ankara University Faculty of Medicine, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boyce MJ, Canning CG, Mahant N, Morris J, Latimer J, Fung VS. Active exercise for individuals with cervical dystonia: a pilot randomized controlled trial. Clin Rehabil. 2013 Mar;27(3):226-35. doi: 10.1177/0269215512456221. Epub 2012 Aug 17. PMID 22904115
- [Background] Barnea ER, MacLusky NJ, DeCherney AH, Naftolin F. Monoamine oxidase activity in the term human placenta. Am J Perinatol. 1986 Jul;3(3):219-24. doi: 10.1055/s-2007-999871. PMID 3718643
- [Background] Mak MK, Wong-Yu IS, Shen X, Chung CL. Long-term effects of exercise and physical therapy in people with Parkinson disease. Nat Rev Neurol. 2017 Nov;13(11):689-703. doi: 10.1038/nrneurol.2017.128. Epub 2017 Oct 13. PMID 29027544
- [Background] Turkish Journal of Neurology 2014; 20: Special Issue 1:34-7
- [Background] Fırat Medical Journal/Firat Med J 2018; 23 (1): 36-38
- [Background] Ceylan, D. (2018). Evaluation of anxiety and depression, cognitive functions and quality of life among non-motor findings in patients followed up with the diagnosis of cervical dystonia and treated with botulinum toxin and their relatives. Unpublished dissertation. Uludag University Faculty of Medicine.
- [Background] Johnson AM, Jimenez-Pardo J, Jenkins ME, Holmes JD, Burke SM. Self-reported physical activity among individuals with Parkinson's disease. Sage Open. (2018) 8:215824401877809. doi: 10.1177/2158244018778096
- [Background] The Effect of Six-Week Physiotherapy and Rehabilitation Program on Balance, Mobility and Quality of Life in a Case with Cervical Dystonia. Fırat Tip Journal 23.1 (2018).
- [Background] De Pauw J, Van der Velden K, Meirte J, Van Daele U, Truijen S, Cras P, Mercelis R, De Hertogh W. The effectiveness of physiotherapy for cervical dystonia: a systematic literature review. J Neurol. 2014 Oct;261(10):1857-65. doi: 10.1007/s00415-013-7220-8. Epub 2014 Jan 12. PMID 24413637